CLINICAL TRIAL: NCT03248596
Title: Interest in Evaluating Primary Hemostasis in Patients With Veno-venous Extracorporeal Membrane Oxygenation (ECMO)
Acronym: ECMO PFA-100
Status: Terminated | Type: Observational
Why Stopped: Obsolete study
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_3023_ECMO PFA-100
Record Dates: First submitted 2017-08-09; First posted 2017-08-14 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Patients With ECMO
Keywords: Extracorporeal Membrane Oxygenation (ECMO); Primary hemostasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is a better understanding of hemorrhagic events causes in patients with ECMO, prevent them and decrease the number of transfusion.

DETAILED DESCRIPTION:
The most frequent complication during ECMO is hemorrhage especially as a curative anticoagulant treatment is necessary. The primary hemostasis is also affected with a von Willebrand disease and thrombopathy, well known but not studied by recent tests.The identification of primary haemostasis deficits with these tools would allow to supply them and decrease the morbi-mortality related to the transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years old
* Patient with ECMO
* Patient hospitalized in an intensive care unit at the University Hospital of Rennes

Exclusion Criteria:

* Known history for constitutional pathology of the primary haemostasis
* Platelets < 100000 / mm3 or hematocrit < 28 % between H+12 and H+24

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with ECMO
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Evaluate primary hemostasis in patient with ECMO at University Hospital of Rennes | Day 5

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France